CLINICAL TRIAL: NCT05861193
Title: Treatment of NCCL Asociated With Gingival Recession With B.O.P.T. Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UV-INV_ETICA-2404840
Record Dates: First submitted 2023-02-28; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-02

CONDITIONS: Abfraction
Keywords: NCCL; B.O.P.T.; Gingival recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cases (Experimental): Patients belonging to the intervention group presented abfraction lesions in upper and/or lower premolars. These abfraction lesions consist of a loss of dental hard tissue at the cervical level of more than 1 mm, and are associated with type 1 gingival recession of the Cairo classification.
  Interventions: Procedure: Treatment of the abfraction with BOPT technique

INTERVENTIONS:
Procedure: Treatment of the abfraction with BOPT technique — The steps to follow for the treatment of abfraction using composite resin and the B.O.P.T. technique will consist of:
  * Selection of the color of the composite, placement of the retraction cord and chamfering of the coronal margin of the lesion;
  * Application of 37% phosphoric acid etching and adhesive in 3 steps; placement of the composite by layers, following the conventional obturation technique.
  * Execution of an overfilling with the composite at the level of the cervical emergence profile of the tooth, with the aim of emphasizing said anatomical particularity.
  * Removal of the retraction cord.
  * Diamond milling with red rim flame diamond bur and contra-angle, positioned from the most apical point of the restoration at an angle of 45º without touching the restored dental portion, with the aim of performing a level rotary gingival curettage from the margin of the restoration.
  * Polishing with a fine-grain flame bur, and polishing discs of decreasing granulometry.

SUMMARY:
The purpose of this clinical trial is to evaluate the gingival margin changes resulting from the treatment with biologically oriented preparation technique (B.O.P.T.) of non-carious cervical lesions (NCCL). In particular, the quantification of the cervical margin is carried out by an intraoral scanning device, both in length and width.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age, all sex;
* Presence of a non-carious lesion with loss of dental hard tissue, located in the cervical third of the tooth, and associated with R1 Cairo dental recession; as well, the tooth must be in a healthy condition.

Exclusion Criteria:

* In the tooth to be treated: presence of tartar, periodontal pocket, gingival hypertrophy and/or dental mobility grades II and III; as well as presence of necrosis, fractures and prosthetic restorations;
* Presence of diabetes, coagulopathies, hemostatic and hormonal alterations, smoking habit of more than 10 cigarettes/day;
* Patients being treated with drugs whose side effects may cause gingival hypertrophy (eg hydantoins);
* Presence of any physical and/or mental condition that prevents voluntary giving informed consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
On the tooth to be treated: Measurement of gingival recession associated to abfraction (before/after treatment). | The initial scan is performed prior to treatment, lasting approximately 5 minutes (maximum). The final scan is performed three month after treatment, once the gingival tissues have healed.
  The gingival recession associated with the abfraction lesion is digitally measured (in mm) through intraoral scanning of the same. Gingival recession is measured from the most coronal portion of the gingival margin to the cementoenamel junction at 3 fixed points (in mesial, medial, and distal).
  A software allows to overlay the initial scan with the post treatment scan; thus, the changes obtained thanks to the treatment in the height of the gingival margin are objectively measured.
On the tooth to be treated: Measurement of the volume of gingiva at the level of the gingival margin (before/after treatment). | The initial scan is performed prior to treatment, lasting approximately 5 minutes (maximum). The final scan is performed three month after treatment, once the gingival tissues have healed.
  The volume of the gingival tissue at the level of the margin, is measured through an initial intraoral scan, at 3 fixed points (the same points measured in the gingival recession, see outcome 1), from the outermost part of the gingiva to the outermost portion of the tooth root, seen in an occlusal view.
  A software allows to overlay the initial scan with the post treatment scan; thus, the volumetric changes obtained thanks to the treatment in the gingival margin are objectively measured.

SECONDARY OUTCOMES:
Periodontal probing of all teeth | Before and after 3 months post-treatment
  Value measured with a Williams periodontal probe with markings at 1-2-3-5-7-8-9-10 mm, from the bottom of the gingival sulcus to the gingival margin at 3 points (mesial, medial and distal).

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Agustin Panadero, PDI-Titular, Principal Investigator — University of Valencia
Locations (1):
- Universidad de Valencia, Valencia, Spain